CLINICAL TRIAL: NCT03744858
Title: The Role of Pyroptosis in Chronic Venous Disease and Its Pathophysiological Implication
Brief Title: The Role of Pyroptosis in Chronic Venous Disease
Acronym: PYROCVD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Clinical Professor, University of Catanzaro
Other Study IDs: ER.CZ.2018.06
Record Dates: First submitted 2018-11-12; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Inflammation; Veins; Complication; Varicose Veins; Varicose Ulcer
Keywords: chronic vein disease; inflammation; pyroptosis
MeSH Terms: conditions — Inflammation; Varicose Veins; Varicose Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A - Participants with CVD: Patients with chronic venous disease (CVD) will undergo peripheral blood draw. Markers of pyroptosis (NETs, Caspase-1 and Cytokines) will be evaluated in blood samples.
  Interventions: Procedure: Peripheral blood draw
- Group B - Healthy Participants: Voluntary healthy subjects will undergo peripheral blood draw. Markers of pyroptosis (NETs, Caspase-1 and Cytokines) will be evaluated in blood samples.
  Interventions: Procedure: Peripheral blood draw

INTERVENTIONS:
Procedure: Peripheral blood draw — Peripheral vein blood draw will be performed to all participants in order to collect blood samples to be evaluated.

SUMMARY:
Enrollment criteria and clinical data collection: following the principles of medical ethics, the development of inclusion and exclusion criteria. Selecting 200 cases of chronic venous disease (CVD) according to the Comprehensive Classification System for Chronic Venous Disorders (CEAP) divided into 6 Clinical stages (C1-C6) (Group A). Selecting 200 healthy participants without CVD (C0) as controls (Group B). Blood samples will be collected from both groups. Markers of pyroptosis (NETs, Caspase-1 and Cytokines) will be evaluated between the two groups and between the subgroups, according to clinical stage, in group A.

DETAILED DESCRIPTION:
Pyroptosis is a pro-inflammatory form of regulated cell death and is dependent on networks of extracellular fibers (NET,s), on the enzymatic activity of inflammatory proteases that belong to the family of cysteine-dependent aspartate-specific proteases (caspase), and cytokines. The role of inflammation has been previously demonstrated in chronic venous disease (CVD), which is a condition that affects up to 80% of adult population in western countries.

According to the Comprehensive Classification System for Chronic Venous Disorders (CEAP) divided into 6 Clinical stages:

C0: no visible or palpable signs of venous disease. C1: telangiectasies or reticular veins. C2: varicose veins. C3: edema. C4a: pigmentation and eczema. C4b: lipodermatosclerosis and atrophie blanche. C5: healed venous ulcer. C6: active venous ulcer.

The aim of this study is to evaluate the role of pyroptosis in the onset and progression of CVD.

The Investigators will select 200 participants with chronic venous disease (CVD) according to Clinical stage of CEAP (C1-C6 patients) [Group A] . The investigators will also select 200 healthy participants without CVD (C0) as controls [Group B].

Peripheral vein blood samples will be collected from both groups. Markers of pyroptosis (NETs, Caspase-1 and Cytokines) will be evaluated between the two groups and between the subgroups of group A, according to clinical stage.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Venous Disease (C1-C6 CEAP classification )

Exclusion Criteria:

* Peripheral artery disease
* Malignant Tumors
* Severe cardiovascular and cerebrovascular disease
* Liver and kidney failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic venous disease (CVD) according clinical stages of CEAP classification:
  C0: no visible or palpable signs of venous disease. C1: telangiectasies or reticular veins. C2: varicose veins. C3: edema. C4a: pigmentation and eczema. C4b: lipodermatosclerosis and atrophie blanche. C5: healed venous ulcer. C6: active venous ulcer.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-11-12 (Estimated); Study Completion 2020-11-12 (Estimated)

PRIMARY OUTCOMES:
Pyroptosis evaluation 1 | 2 years
  NETs evaluation to be presented in ng/ml
Pyroptosis evaluation 2 | 2 years
  Caspase-1 evaluation to be presented in pg/ml
Pyroptosis evaluation 3 | 2 years
  IL-1 β, IL-4, IL-10, IL-18, and TNF-α evaluation to presented in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Serra, MD, PhD, Principal Investigator — University Magna Graecia of Catanzaro
Locations (1):
- CIFL- Interuniversity Center of Phlebolymphology, Catanzaro, Italy